CLINICAL TRIAL: NCT06983561
Title: An Exploratory and Proof of Concept Study to Characterize and Describe the Population of Subjects Suffering From Moderate to Severe Atopic Dermatitis, Treated and Controlled by Systemic Treatments and Their Needs and Expectations Regarding the Use of Emollient
Brief Title: Description of the Population With Moderate to Severe Atopic Dermatitis, Treated by Systemic Treatments and Needs Regarding Emollients
Status: Recruiting | Type: Observational
Sponsor: Pierre Fabre Dermo Cosmetique (Industry)
Responsible Party: Sponsor
Other Study IDs: ADNEEDS
Record Dates: First submitted 2025-05-12; First posted 2025-05-21 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Subject with atopic dermatitis

SUMMARY:
Atopic dermatitis (AD) is a common chronic inflammatory skin disease, affecting both children (15- 20%) and adults (2-5%). The pathogenesis of AD is complex and multifactorial, including skin barrier dysfunction and immune dysregulation. AD often requires a long management and has a major impact on quality of life. For mild to moderate disease, first-line treatment involves topical therapies including corticosteroids and calcineurin inhibitors. Patients with more severe and refractory symptoms require systemic treatments as phototherapy, conventional systemic treatments (cyclosporine, methotrexate…), biologics and JAK-inhibitors.

Regardless of the severity of the disease, additional basic topical treatment with emollient is the mainstay of the management. Emollients, commonly referred to as moisturizing creams are well known for their role in moisture retention, barrier repair and symptom control in AD.

Publications on emollient in atopic dermatitis are numerous but there are limited data on how patients with AD treated by systemic treatment use and evaluate emollients.

The aim of this study is to characterize and describe the population of subjects suffering from moderate to severe AD, treated and controlled by systemic treatments in terms of pathology, the state of their skin at this stage of their systemic treatment (controlled period), their habits, needs and expectations regarding the use of emollient.

This study will be conducted as an exploratory, proof of concept, international, multicentric study in adult subjects suffering from moderate to severe AD, treated and controlled by systemic treatments.

2 visits are planned: Visit 1 (Day 1): Inclusion Visit 2 (from Day 2 to Day 8): End-of-study visit - remote visit for subject's questionnaire filling The maximal duration of participation for a subject is 8 days.

ELIGIBILITY:
Inclusion Criteria:

Criteria related to the population:

* Subject aged between 18 and 75 years included
* Subject having signed his/her written informed consent for his/her participation in the study
* Subject affiliated to a social security system or health insurance, or is a beneficiary (if required by national regulations
* Subject with appropriate hardware (smartphone and/or tablet and/or computer) to complete digital questionnaires
* Subject with a mailbox and internet access to create his account to complete digital questionnaires

Criteria related to the disease and treatment:

• Subject with moderate to severe atopic dermatitis controlled by systemic treatment, meaning:

* Using systemic treatment for atopic dermatitis (biologics, janus kinase inhibitors or conventional immunosuppressants) initiated for at least 6 months at the time of the inclusion visit
* With an unchanged systemic treatment dose for at least 2 months at the time of the inclusion visit,
* And with an vIGA-ADTM ≤ 2 (Mild).

Non Inclusion criteria:

Criteria related to the population:

* Subject unable to understand the information given including study procedures (for linguistic or psychiatric reasons) and to give his/her consent in writing and to report required information in writing in the questionnaire
* For woman of childbearing potential: pregnant or breastfeeding or planning to be pregnant during the study
* Subject who has forfeited his/her freedom by administrative or legal award or is under guardianship
* Subject who, in the judgement of the investigator, is not likely to be compliant with study-related constraints and requirements
* Subject who is currently participating, who plans to participate or who has participated within the previous weeks or months in another clinical study liable to interfere with the study assessments according to the investigator's assessment
* Subject is in a position likely to represent a conflict of interest and/or is a family member of any people involved in the conduct of the study (secretary, nurse, technician,…), of the investigational site

Criteria related to the diseases / skin condition:

• Subject having a dermatological condition, an acute, chronic or progressive disease or history of disease liable to interfere with the study data or considered by the Investigator hazardous for the subject or incompatible with the study requirements

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects will be enrolled from the investigator's outpatients reception and/or from the database of the centre.
  The subjects corresponding to eligibility criteria may receive a phone call, a letter or an e-mail proposing to participate to the clinical study.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-06-16 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
Epidemiological data | Visit 2 (from Day 2 to Day 8)
  By a questionnaire filled in by all subjects to characterize and describe the population in terms of pathology, state of the skin, habits, needs and expectations of patients regarding the use of emollient

CONTACTS AND LOCATIONS:
Locations (1):
- Allergologie et Immunologie Clinique, CHU Lyon Sud, Pierre-Bénite, France